CLINICAL TRIAL: NCT00416039
Title: Clinical Randomized Study of Sublingual Midazolam in Association With Morphine by Oral Route in Arm Fracture in Children at the Emergency Children Care
Brief Title: Efficacy of Sublingual Midazolam in Association With Oral Morphine in Children Analgesia After Bone Fracture
Acronym: MIDAZODOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P051033
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Fractures
Keywords: midazolam; sublingual; oral morphine; children; bone fracture; bone fracture with a deformed member
MeSH Terms: conditions — Fractures, Bone | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Midazolam and morphine
  Interventions: Drug: Midazolam
- 2 (Placebo Comparator): placebo, Nacl 0.9 %, morphine 0.5 mg/kg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midazolam — 0.2 mg/kg of sublingual midazolam and 0.5 mg/kg of morphine
  Arms: 1
Drug: Placebo — placebo at 0.2 mg/kg and morphine 0.5 mg/kg
  Arms: 2

SUMMARY:
It is a randomized simple-blind monocentric study; the group A will receive oral morphine with placebo and the group B will receive oral morphine with sublingual midazolam. The aim of this study is to show a more important pain decrease in the group taking midazolam versus placebo.

DETAILED DESCRIPTION:
Fracture is often responsible of pain in the paediatric emergency department (ED). This pain is very severe and needs effective drugs.

During a study made at the ED of Necker Enfants Malades Hospital, it has been shown that the oral morphine had a limited action on this kind of pain. Therefore it is interesting to increase the analgesia by making a drug association, for example with the midazolam witch is a benzodiazepine with a sedative and anxiolytic action, and which has got the MMA for the intravenous and the intra rectal forms for children older than 6 months.

The intravenous form has some disadvantages like an extra work and an increase of risk of side effects.

That is why the sublingual form seems to be interesting in this context. Even if some studies have shown the benefit of midazolam as a preanesthetic medication given to children scheduled for a surgical procedure, none has shown the interest of sublingual midazolam associated with oral morphine to relieve the pain due to a displaced fracture.

The aim of this study is to show a more important pain decrease in the group taking midazolam versus placebo.

It is a randomized simple-blind monocentric study; the group A will receive oral morphine with placebo and the group B will receive oral morphine with sublingual midazolam . The pain will be quantified thanks to the visual analogical scale (VAS)before and 30 minutes after the drugs administration, and we will try to show a difference of 15 points(on 100) of the VAS at 30 minutes between the two groups.

60 patients aged from 5 to 16 years old and having a displaced fracture will be enrolled in this study which will last 1 year.

Patients having a contra-indication for morphine and midazolam won't be enrolled as patients with femoral fracture which needs a local anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* children between 5 and 16 years old
* children with a disjoined bone fracture
* children needed oral morphine analgesia
* written informed consent from one or the two parents or legal pad

Exclusion Criteria:

* ASA score > 2
* concomitant administration of oral analgesia (level II WHO classification) less than 6 hours
* concomitant administration of benzodiazepine less than 24 hours

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Difference in the measurement of pain analogical scale values at 30 minutes between the two groups | after administration until 120 minutes

SECONDARY OUTCOMES:
Pain Analogical scale Values at 15, 30 minutes, 1 hour, 1h30 and 2 hours. | after administration until 120 minutes
Pain Analogical scale Values after the treatment of the fracture | after administration until 120 minutes
Respiratory rate, Oxymetry | after administration until 120 minutes
Conscience (lethargy or irritability) | after administration until 120 minutes
nausea, | after administration until 120 minutes
skin hyperesthesia, rash | after administration until 120 minutes
children cooperation | after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gérard CHERON, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Necker enfants Malade - Department of Pediatric Emergency, Paris, France

REFERENCES:
- [Background] 21480984
- [Result] Wille-Ledon C, Chappuy H, Giraud C, Treluyer JM, Cheron G. Comparison of a morphine and midazolam combination with morphine alone for paediatric displaced fractures: a randomized study. Acta Paediatr. 2011 Nov;100(11):e203-7. doi: 10.1111/j.1651-2227.2011.02311.x. Epub 2011 May 11. PMID 21480984